CLINICAL TRIAL: NCT06216886
Title: Randomized Controlled Trial of Intradermal Injections of OnabotulinumtoxinA vs Saline for Trigeminal Neuralgia.
Brief Title: OnabotulinumtoxinA for Trigeminal Neuralgia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Meredith Barad, Clinical Associate Professor of Anesthesiology (Pain) and Neurology & Neurological Sciences, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 66036
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Trigeminal Neuralgia
Keywords: botox; injection; trigeminal neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — Botulinum Toxins, Type A; Sodium Chloride; Injections

STUDY DESIGN:
Intervention Model Description: This will be a randomized controlled trial of onabotulinumtoxinA versus Saline intradermal injections into the affected trigeminal distributions. The RCT will be enriched with all participants being initial responders to a preliminary round of onatbotulinumtoxinA.
Who Masked: Participant, Care Provider, Investigator
Masking Description: After the initial round of botox, all participants will be randomized to either onabotA or saline. The randomization will performed by a provider who is not a care provider or proceduralist.
  The patient will be blinded, the proceduralist will be blinded and the care provider will be blinded. Data will be stored and not reviewed by research team until the study closes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- OnabotulinumtoxinA (Experimental): Intradermal injections will be placed in the affected trigeminal territories according to a specific facial map that we have developed.
  Interventions: Drug: OnabotulinumtoxinA 100 UNT [Botox]
- Saline (Placebo Comparator): The same procedure will be followed as above, but saline will be injected instead of onabotA
  Interventions: Drug: Sodium Chloride 0.9% for Injection, Preservative Free

INTERVENTIONS:
Drug: OnabotulinumtoxinA 100 UNT [Botox] — Intradermal injections will be placed in 25 unit aliquots allocated per affected trigeminal distribution. For example, if the target is the V1 territory, then the patient would get 25 units injected into the V1 distribution. This would be divided into 2.5 units per injection in 10 injection sites as outlined on the map. If V1/V2 were affected, the patient would get 50 units of onabotA. Maximum dose of 75 units if all three trigeminal distributions are involved. We have developed a specific map for administering the doses and this will be followed.
  Other Names: Botox
  Arms: OnabotulinumtoxinA
Drug: Sodium Chloride 0.9% for Injection, Preservative Free — intradermal injections will be placed in 25 unit aliquots allocated per affected trigeminal distribution. For example, if the target is the V1 territory, then the patient would get 25 units injected into the V1 distribution. This would be divided into 2.5 units per injection in 10 injection sites as outlined on the map. If V1/V2 were affected, the patient would get 50 units of saline. Maximum dose of 75 units if all three trigeminal distributions are involved. We have developed a specific map for administering the doses and this will be followed.
  Other Names: Saline
  Arms: Saline

SUMMARY:
A randomized controlled trial comparing Onabotulinumtoxin A to saline (placebo) for Trigeminal Neuralgia.

DETAILED DESCRIPTION:
This study will offer onabotulinumtoxin A (Botox) delivered intradermally into the region of pain for the patient with trigeminal neuralgia. Should they derive benefit from the procedure (as determined by decrease in the frequency of attacks), then they will be randomized to receive either onabotulinumtoxin A or saline and followed for 3 months. This study hopes to provide strong data that this is a treatment option for patients with TN who have failed medications, but are not ready for or do not want to undergo surgery.

ELIGIBILITY:
Inclusion Criteria:

Men and women age 18 or older

* Judged to be of legal competence
* Sufficient knowledge of written and spoken English
* Capable of attending regular in-person visits
* Have failed/not a candidate/do not want surgery
* Inadequate response to medication - at least 2 trials
* Meeting ICHD criteria for Classical Trigeminal Neuralgia 13.1.1.1
* Patients with frequency > 10 attacks per week
* Stable dose of medications in the last 2 weeks

Exclusion Criteria:

* Secondary or Idiopathic TN, or Painful Trigeminal Neuropathy as defined by the ICHD (13.1.1.2, 13.1.1.3, 13.1.2)
* Pregnant or breast feeding (while it is rare that a patient will be pregnant with TN, there is not sufficient data to say definitively that onabotA is ok to use during pregnancy and nursing, it is still rated Class C)
* Neuromuscular disease
* On aminoglyocosides
* Not currently enrolled in any other studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Number of TN Attacks per week | compare data from week -1(7 days prior to starting study) and week 4(7 days during the 4th week after treatment))
  Frequency of TN attacks before and after onabotA injection over a seven day period

SECONDARY OUTCOMES:
Change in PROMIS Computer Adaptive Tests (PROMIS PROFILE CAT V1.0 -29) | compare data from week -1(7 days prior to starting study) and week 4(7 days during the 4th week after treatment)
  Computer adaptive tests (CATs) assess anxiety, depression, fatigue, pain interference, physical function, sleep disturbance and ability to participate in social roles and activities, and pain intensity.
Change in Severity of Attacks Based using the numerical rating scale (NRS) | compare data from week -1(7 days prior to starting study) and week 4(7 days during the 4th week after treatment)
  Average severity of attack over a 7 day period
Change In Baseline Pain Average using the numerical rating scale (NRS) | compare data from week -1(7 days prior to starting study) and week 4(7 days during the 4th week after treatment)
  baseline pain average over a seven day period
Change In Acute Medication Use | compare data from week -1(7 days prior to starting study) and week 4(7 days during the 4th week after treatment)
  Number of doses of any acute medication use over a 7 day period
Change In Patient Global Impression of Change | week 4
  A single self administered question given at week 4

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Barad, MD, Principal Investigator — Stanford University
Locations (1):
- Meredith Barad, Stanford, California, United States

REFERENCES:
- [Background] undefined
- [Background] Morra ME, Elgebaly A, Elmaraezy A, Khalil AM, Altibi AM, Vu TL, Mostafa MR, Huy NT, Hirayama K. Therapeutic efficacy and safety of Botulinum Toxin A Therapy in Trigeminal Neuralgia: a systematic review and meta-analysis of randomized controlled trials. J Headache Pain. 2016 Dec;17(1):63. doi: 10.1186/s10194-016-0651-8. Epub 2016 Jul 5. PMID 27377706
- [Background] Wei J, Zhu X, Yang G, Shen J, Xie P, Zuo X, Xia L, Han Q, Zhao Y. The efficacy and safety of botulinum toxin type A in treatment of trigeminal neuralgia and peripheral neuropathic pain: A meta-analysis of randomized controlled trials. Brain Behav. 2019 Oct;9(10):e01409. doi: 10.1002/brb3.1409. Epub 2019 Sep 21. PMID 31541518
- [Background] Hu Y, Guan X, Fan L, Li M, Liao Y, Nie Z, Jin L. Therapeutic efficacy and safety of botulinum toxin type A in trigeminal neuralgia: a systematic review. J Headache Pain. 2013 Aug 21;14(1):72. doi: 10.1186/1129-2377-14-72. PMID 23964790
- [Background] Li S, Lian YJ, Chen Y, Zhang HF, Ma YQ, He CH, Wu CJ, Xie NC, Zheng YK, Zhang Y. Therapeutic effect of Botulinum toxin-A in 88 patients with trigeminal neuralgia with 14-month follow-up. J Headache Pain. 2014 Jun 22;15(1):43. doi: 10.1186/1129-2377-15-43. PMID 24952600
- [Background] Zuniga C, Piedimonte F, Diaz S, Micheli F. Acute treatment of trigeminal neuralgia with onabotulinum toxin A. Clin Neuropharmacol. 2013 Sep-Oct;36(5):146-50. doi: 10.1097/WNF.0b013e31829cb60e. PMID 24045604
- [Background] Zhang H, Lian Y, Ma Y, Chen Y, He C, Xie N, Wu C. Two doses of botulinum toxin type A for the treatment of trigeminal neuralgia: observation of therapeutic effect from a randomized, double-blind, placebo-controlled trial. J Headache Pain. 2014 Sep 27;15(1):65. doi: 10.1186/1129-2377-15-65. PMID 25263254
- [Background] Shehata HS, El-Tamawy MS, Shalaby NM, Ramzy G. Botulinum toxin-type A: could it be an effective treatment option in intractable trigeminal neuralgia? J Headache Pain. 2013 Nov 19;14(1):92. doi: 10.1186/1129-2377-14-92. PMID 24251833
- [Background] Tangney T, Heydari ES, Sheldon BL, Shetty A, Argoff CE, Khazen O, Pilitsis JG. Botulinum Toxin as an Effective Treatment for Trigeminal Neuralgia in Surgical Practices. Stereotact Funct Neurosurg. 2022;100(5-6):314-320. doi: 10.1159/000526053. Epub 2022 Aug 9. PMID 35944492
- See also: NIH PROMIS MEASURES — https://www.healthmeasures.net/explore-measurement-systems/promis
- See also: Quality of Life Scale instructions and References — https://resourcelibrary.stfm.org/viewdocument/quality-of-life-scale-qols?CommunityKey=2751b51d-483f-45e2-81de-4faced0a290a&tab=librarydocuments